CLINICAL TRIAL: NCT07303543
Title: Preventing Muscle Loss in the Early Postoperative Period of Bariatric Surgery With a Combination of Whey Protein, Hydrolyzed Collagen, and Resistance Exercise: A Prospective, Randomized, Controlled Clinical Study
Brief Title: Preventing Muscle Loss After Bariatric Surgery: Protein-Collagen Supplementation and Resistance Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Rüken Aslınur Samanci, Lecturer, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E-66291034-772.02-3053
Record Dates: First submitted 2025-11-17; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Bariatric Surgery; Muscle Loss
Keywords: Bariatric Surgery; Collagen; Resistance exercise; Whey protein; Muscle loss
MeSH Terms: conditions — Muscular Atrophy | interventions — Vitamins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (CG) (Active Comparator): Whey protein supplementation will be provided. Vitamin and mineral supplementation will be administered. No resistance exercise will be performed. Participants will follow bariatric surgery nutrition guidelines and maintain their regular physical activities.
  A comparison will be made with the other groups as the control group.
  Interventions: Dietary Supplement: Whey protein supplement; Dietary Supplement: Vitamin and Mineral Supplementation
- Whey Protein + Collagen + Exercise Group (WPCEG) (Experimental): Collagen-containing whey protein supplementation will be provided. Vitamin and mineral supplementation will be given. Resistance exercises will be performed. Participants will follow bariatric surgery nutrition guidelines and maintain their physical activities.
  They will begin the resistance exercise program in the 4th week after surgery.
  Interventions: Dietary Supplement: Whey protein supplement; Dietary Supplement: Hydrolyzed Collagen Supplement; Dietary Supplement: Vitamin and Mineral Supplementation; Behavioral: Resistance Exercise Program
- Whey Protein + Collagen + Non-Exercise Group (WPCG) (Experimental): Collagen-containing whey protein supplementation will be provided. Vitamin and mineral supplementation will be administered. No resistance exercises will be performed. Participants will follow bariatric surgery nutrition guidelines and maintain their physical activities.
  Interventions: Dietary Supplement: Whey protein supplement; Dietary Supplement: Vitamin and Mineral Supplementation
- Whey Protein + Exercise Group (WPEG) (Experimental): Whey protein supplementation will be provided. Vitamin and mineral supplementation will be given. Resistance exercises will be performed. Participants will follow bariatric surgery nutrition guidelines and maintain their physical activities.
  They will begin the resistance exercise program in the 4th week after surgery.
  Interventions: Dietary Supplement: Whey protein supplement; Dietary Supplement: Vitamin and Mineral Supplementation; Behavioral: Resistance Exercise Program

INTERVENTIONS:
Dietary Supplement: Whey protein supplement — Oral whey protein supplement provided daily according to bariatric surgery nutrition protocol.
Dietary Supplement: Hydrolyzed Collagen Supplement — Oral hydrolyzed collagen supplement provided daily in combination with whey protein.
  Arms: Whey Protein + Collagen + Exercise Group (WPCEG)
Dietary Supplement: Vitamin and Mineral Supplementation — Routine vitamin and mineral supplementation according to bariatric surgery follow-up protocol.
Behavioral: Resistance Exercise Program — Structured resistance exercise program initiated at postoperative week 4, supervised, 3 times per week.
  Arms: Whey Protein + Collagen + Exercise Group (WPCEG); Whey Protein + Exercise Group (WPEG)

SUMMARY:
The aim of this clinical trial is to investigate the effectiveness of collagen, considered a new approach to prevent muscle mass loss after bariatric surgery, and to demonstrate the relationship between this effect and exercise. The key questions it aims to answer are:

Does whey protein supplementation with collagen combined with resistance exercise prevent muscle mass loss after bariatric surgery? Do whey protein supplementation with collagen combined with resistance exercise affect fat mass after bariatric surgery?

Researchers will compare collagen with whey protein.

The study groups and interventions to be implemented are summarized below:

Group 1: Control Group (CG; n: 10) Whey protein supplementation will be administered Vitamin and mineral supplementation will be administered No resistance exercise will be performed The participants will eat according to bariatric surgery nutrition guidelines and perform physical activities.

Group 2: Whey Protein + Collagen + Exercise Group (WPCEG; n: 10) Whey protein supplements with collagen will be given. Vitamin and mineral supplements will be given. Resistance exercise will be performed. They will eat according to bariatric surgery nutrition guidelines and perform physical activities.

They will begin a resistance exercise program 4 weeks after surgery.

Group 3: Whey Protein + Collagen + No Exercise Group (WPCG; n: 10) Whey protein supplements with collagen will be given. Vitamin and mineral supplements will be given. No resistance exercise will be performed. They will eat according to bariatric surgery nutrition guidelines and perform physical activities.

Group 4: Whey Protein + Exercise Group (WPEG; n: 10) Whey protein supplements will be given. Vitamin and mineral supplements will be given. Resistance exercise will be performed. They will eat according to bariatric surgery nutrition guidelines and perform physical activities.

A resistance exercise program will begin at 4 weeks post-operatively.

DETAILED DESCRIPTION:
Bariatric surgery is an effective method for treating obesity, but a significant decrease in skeletal muscle mass can be observed in the early postoperative period. This loss of muscle mass can negatively affect physical functions, reduce metabolic rate, and make long-term weight maintenance more difficult. Therefore, developing strategies to prevent muscle loss after bariatric surgery is of great clinical importance.

The use of whey protein to support muscle protein synthesis in the postoperative period is a common practice. In recent years, there has been increased scientific interest in the potential of collagen peptides, especially when used in conjunction with resistance exercise, to contribute to muscle mass preservation. However, studies evaluating the combined effect of collagen supplementation and exercise programs in addition to whey protein in individuals undergoing bariatric surgery are limited.

This clinical study aims to investigate the effectiveness of adding collagen to standard whey protein supplementation and a resistance exercise program in preventing muscle loss. Four different groups will be designed to evaluate the independent and combined effects of collagen and exercise:

1. Group receiving only whey protein,
2. Whey + collagen + exercise group,
3. Whey + collagen but no exercise group,
4. Whey + exercise but no collagen group.

All participants will follow a standard post-bariatric surgery nutrition protocol and receive routine vitamin and mineral supplements. The resistance exercise program will begin four weeks after surgery; it will consist of progressively more intense, supervised exercises targeting large muscle groups. Body composition assessments will be performed at baseline and at specified follow-up weeks. The primary outcome measure is change in skeletal muscle mass; secondary outcome measures are fat mass, functional capacity, and exercise compliance.

This study is expected to contribute to the identification of optimal nutrition and exercise strategies to reduce muscle loss after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Being between 20-50 years old
* Body mass index; 35 ≤ BMI< 60 kg/m2
* Not being pregnant
* Not being addicted to alcohol and drugs
* Not having entered menopause
* No exercise restrictions

Exclusion Criteria:

* Having at least one of the following inflammatory bowel diseases, upper gastrointestinal bleeding, advanced psychiatric diseases, cancer, and kidney failure.
* using statins
* be pregnant
* Being addicted to alcohol and drugs
* to have entered menopause
* Having exercise restrictions
* Becoming a professional athlete
* Having done more than 60 minutes of regular and structured exercise per week in the last year

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — man and woman
Enrollment: 35 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in Skeletal Muscle Mass (kg) Measured by BIA | Baseline (preoperative), postoperative week 4 (day 29), and postoperative week 12 (day 85)
  Skeletal muscle mass (kg) will be measured using a multi-frequency bioelectrical impedance analysis (BIA) device. The outcome will be reported as the mean change from baseline at each time point in each study group.

SECONDARY OUTCOMES:
Change in Fat Mass (kg) Measured by BIA | Baseline, week 4, and week 12
  Fat mass (kg) will be measured using BIA. Results will be summarized as the mean change from baseline for each group.

CONTACTS AND LOCATIONS:
Overall Officials: Halit E Taşkın, Dr., Principal Investigator — Cerrahpaşa Faculty of Medicine, General Surgery; Nihal Z Erdem, PhD, Principal Investigator — Istanbul Medipol University, Nutrition and Dietetics; Bürke Köksalan, PhD, Principal Investigator
Locations (1):
- Istanbul Medipol University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because this study involves identifiable clinical and nutritional data collected at a single center, and participant privacy cannot be fully ensured despite anonymization